CLINICAL TRIAL: NCT00648674
Title: A Prospective, Single-Site Study to Identify and Characterize the Molecular Mechanisms of Apligraf in Non-healing Wounds of Subjects With Venous Leg Ulcers
Brief Title: A Post-Marketing Clinical Study of Apligraf for Venous Leg Ulcers
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Organogenesis (Industry)
Responsible Party: Damien Bates, MD, PhD, Chief Medical Officer, Organogenesis Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-MOA-001-AG
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Varicose Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Apligraf
  Interventions: Device: Apligraf

INTERVENTIONS:
Device: Apligraf — Applied at Day 0, possible re-application at Week 6

SUMMARY:
Single site clinical study utilizing the novel technology of microarrays to identify and characterize the molecular mechanisms through which Apligraf promotes healing of venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Subject has non-infected partial or full-thickness venous leg ulcer for a duration of four weeks or greater which has not adequately responded to conventional therapy
* Stage II or III ulcer as defined by the IAET/WOCN ulcer classification guide listed in Appendix IV.
* Subject is female and 18 years of age or older.
* Subject with venous leg ulcer (target ulcer) between 5 - 40 cm2 in size.
* Sexually active females must be practicing a medically proven form of contraception during the course of the study period.
* Subject or legal guardian must have read, understood and signed an institutional review board (IRB) approved Informed Consent Form.
* Subject and/or legal guardian must be able and willing to follow study procedures and instructions.

Exclusion Criteria:

* Subject whose target ulcer has healed 60% or greater in area from post debridement (if applicable) Baseline Screen (Visit 1) to post debridement Day 0 (Visit 2) as determined by wound tracings.
* Subjects who are being treated with VAC® (Vacuum Assisted Closure™) Therapy.
* Subject has arterial disease as determined by an Ankle Brachial Index (ABI ) of <0.65.
* Subject with any systemic condition like uncontrolled diabetes mellitus (glycosylated HbA1C > 12%), cancer (biopsy confirmed active malignancy), positive HIV test, or any disorder(s) that may compromise wound healing.
* Subjects who are currently receiving, or have received at any time within one month prior to entry into the study, corticosteroids (>15 mg/day), immunosuppressive agents, radiation therapy, hemodialysis or chemotherapy. Anticipated use of the above agents will exclude subjects from entry into the study.
* Clinical vasculitis, severe rheumatoid arthritis, and other collagen vascular diseases.
* Signs and symptoms of cellulitis or osteomyelitis.
* Necrotic or avascular ulcer beds.
* Venous leg ulcer with exposed bone, tendon or fascia.
* Subject with the presence of recent infections in the area intended for treatment.
* Known hypersensitivity to bovine collagen or to the components of the Apligraf agarose shipping medium.
* Subject who is lactating or pregnant (hCG positive as determined by lab testing).
* Subject with liver (ALT/SGPT, ALP, AST/SGOT, bilirubin, Albumin, total protein, LDH) and/or renal function (BUN and creatinine) tests greater than 2 x upper limit of normal (ULN) or Albumin < 2.5 mg/dL.
* Subject enrolled in any wound or investigational device study for any disease within the past four weeks.
* Subject previously treated at target site with Apligraf, Dermagraft or any other cell therapy at the target site.
* Subject with a history of alcohol or substance abuse within the previous year, which could interfere with study compliance such as inability to attend scheduled study visits or compliance with home dressing changes.
* Subject who, in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To use the novel technology of microarrays to identify and characterize the molecular mechanisms through which Apligraf promotes healing of venous leg ulcers. | 2 weeks

SECONDARY OUTCOMES:
Determine how venous leg ulcer (VLU) wounds transition from chronic to acute wound healing | 2 weeks
Examine how Apligraf rescues deficiencies of chronic wounds (VLU) and promotes transition from chronic to acute wound | 2 weeks
Determine growth factors induced by Apligraf in the wound | 2 weeks
Determine growth factors suppressed by Apligraf in the wound | 2 weeks
Safety endpoints assessed by monitoring adverse events | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Damien Bates, MD, PhD, FRACS (Plast.), Study Director — Organogenesis Inc.